CLINICAL TRIAL: NCT00086866
Title: Randomized, Open Phase II Study of Immunization With the Recombinant MAGE-3 Protein Combined With Adjuvant AS02B or AS15 in Patients With Unresectable and Progressive Metastatic Cutaneous Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed With Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16032-18031; EORTC-18031; EORTC-16032; GSK-249553/008; 2004-001937-40 (EudraCT Number)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: D1/3-MAGE-3-His fusion protein
Biological: SB-AS02B adjuvant
Biological: SB-AS15 adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase II trial is studying two different regimens of vaccine therapy and comparing them to see how well they work in treating patients with stage III or stage IV melanoma that cannot be removed with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the objective response rate (complete and partial response) in patients with unresectable stage III or stage IV M1a cutaneous melanoma immunized with vaccine comprising D1/3-MAGE-3-His fusion protein and SB-AS02B adjuvant vs SB-AS15 adjuvant.
* Compare the activity of SB-AS02B adjuvant vs SB-AS15 adjuvant, in terms of maximizing the antigenicity of MAGE-3, in patients treated with these regimens.
* Compare the rate of grade 3/4 vaccine-related toxicity in patients treated with these regimens.

Secondary

* Compare progression-free survival in patients treated with these regimens.

OUTLINE: This is a randomized, open label, parallell-group, multicenter study. Patients are stratified according to disease stage (III in transit vs other stage III vs IV), presence of lesion ≥ 20 mm (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Induction therapy

  * Arm I: Patients receive immunization comprising D1/3-MAGE-3-His fusion protein and SB-AS02B adjuvant intramuscularly (IM) once weekly on weeks 1, 3, 5, 7, 9, and 11.
  * Arm II: Patients receive immunization comprising D1/3-MAGE-3-His fusion protein SB-AS15 adjuvant IM once weekly on weeks 1, 3, 5, 7, 9, and 11.

Patients achieving a clinical complete response (CR), partial response (PR), stable disease (SD), or slow progressive disease (SPD) proceed to maintenance therapy.

* Maintenance therapy: Patients in both arms receive immunization (according to their randomized arm) once weekly on weeks 15, 18, 21, 24, 27, 30, 34, 40, 46, and 52.

Patients maintaining a CR, PR, or SD proceed to long-term treatment.

* Long-term treatment: Beginning 3 months after completion of maintenance therapy, patients in both arms receive immunization (according to their randomized arm) once every 3 months for 4 courses and then once every 6 months for 4 courses.

Treatment continues in both arms in the absence of disease progression that does not correspond to SPD status, unacceptable toxicity, or the diagnosis of an autoimmune disease.

Patients are followed every 12 weeks.

PROJECTED ACCRUAL: A total of 68 patients (34 patients per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous melanoma

  * Unresectable stage III OR stage IV M1a disease
* Documented progressive disease within the past 12 weeks
* Measurable disease
* Skin, soft tissue, or lymph node metastasis allowed provided the disease is not amenable to curative treatment with surgery
* Tumor must express the MAGE-3 gene by reverse transcription polymerase chain reaction analysis (more than 1% of the positive MAGE-3 control included in the assay)
* No visceral metastases within the past 56 days by imaging

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ lower limit of normal (LLN)
* WBC ≥ LLN
* Lymphocyte count ≥ LLN
* Platelet count ≥ LLN
* No bleeding disorders

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* Lactic dehydrogenase ≤ ULN
* AST and ALT ≤ 2 times ULN
* PT and aPTT normal
* Hepatitis B surface antigen negative (antibody test may be positive)
* Hepatitis C antibody negative

Renal

* Creatinine ≤ ULN

Cardiovascular

* No clinically significant heart disease (CTC grade III or IV)

Immunologic

* No autoimmune disease (vitiligo allowed)
* No anti-nuclear antibody titer ≥ 1/320 OR equal to 1/160 AND auto-antibodies directed against specific auto-antigens
* No immunodeficiency
* No active infection requiring antibiotic therapy
* HIV negative

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other malignancy within the past 5 years except surgically cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other serious acute or chronic illness requiring concurrent medications
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 8 weeks since prior adjuvant vaccine therapy
* No prior vaccine therapy containing a MAGE-3 antigen
* No prior vaccine therapy for metastatic melanoma
* No concurrent immunomodulating agents (e.g., BCG)

Chemotherapy

* No prior systemic chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* No concurrent corticosteroids

  * Concurrent prednisone or equivalent allowed provided the dose is ≤ 40 mg/day and treatment duration is for no more than 3 weeks
  * Concurrent inhaled and topical steroids are allowed

Radiotherapy

* No prior radiotherapy to the spleen
* No concurrent radiotherapy to > 20% of all existing lesions (i.e., target lesions, non-target lesions, and nonmeasurable lesions)

  * Concurrent local low-dose (≤ 20 Grays) radiotherapy allowed

Surgery

* Recovered from prior surgery or biopsy
* No prior organ allograft
* No prior splenectomy
* Concurrent surgery to a limited number of lesions allowed for patients with a complete response, partial response, or stable disease after at least 3 courses of study therapy

Other

* No prior systemic anticancer therapy
* More than 4 weeks since prior isolated limb perfusion therapy
* No other concurrent anticancer therapy
* No other concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2004-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response and partial response) as assessed by RECIST criteria
Vaccine-related toxicity as assessed by CTCAE v3

SECONDARY OUTCOMES:
Rate of stabilization as assessed by RECIST criteria
Rate of mixed response as assessed by RECIST criteria
Rate of immune response
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Willem H. J. Kruit, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center; Cornelis J. A. Punt, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (21):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
- France (6):
  - Clinique Sainte-Marguerite, Hyères
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Hopital St. Eloi, Montpellier
  - CHR Hotel Dieu, Nantes
  - Institut Curie Hopital, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Klinikum der Stadt Mannheim, Mannheim
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Italy (4):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Universita di Siena, Siena
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Saint Bartholomew's Hospital, London, England
  - Christie Hospital NHS Trust, Manchester, England

REFERENCES:
- [Result] Kruit WH, Suciu S, Dreno B, et al.: Immunization with recombinant MAGE-A3 protein combined with adjuvant systems AS15 or AS02B in patients with unresectable and progressive metastatic cutaneous melanoma: A randomized open-label phase II study of the EORTC Melanoma Group (16032- 18031). [Abstract] J Clin Oncol 26 (Suppl 15): A-9065, 2008.
- [Result] Louahed J, Gruselle O, Gaulis S, et al.: Expression of defined genes identified by pretreatment tumor profiling: association with clinical responses to the GSK MAGE- A3 immunotherapeutic in metastatic melanoma patients (EORTC 16032-18031). [Abstract] J Clin Oncol 26 (Suppl 15): A-9045, 2008.
- [Derived] Kruit WH, Suciu S, Dreno B, Mortier L, Robert C, Chiarion-Sileni V, Maio M, Testori A, Dorval T, Grob JJ, Becker JC, Spatz A, Eggermont AM, Louahed J, Lehmann FF, Brichard VG, Keilholz U. Selection of immunostimulant AS15 for active immunization with MAGE-A3 protein: results of a randomized phase II study of the European Organisation for Research and Treatment of Cancer Melanoma Group in Metastatic Melanoma. J Clin Oncol. 2013 Jul 1;31(19):2413-20. doi: 10.1200/JCO.2012.43.7111. Epub 2013 May 28. PMID 23715572
- [Derived] Ulloa-Montoya F, Louahed J, Dizier B, Gruselle O, Spiessens B, Lehmann FF, Suciu S, Kruit WH, Eggermont AM, Vansteenkiste J, Brichard VG. Predictive gene signature in MAGE-A3 antigen-specific cancer immunotherapy. J Clin Oncol. 2013 Jul 1;31(19):2388-95. doi: 10.1200/JCO.2012.44.3762. Epub 2013 May 28. PMID 23715562